CLINICAL TRIAL: NCT06281548
Title: Determining the Feasibility and Acceptability of a Novel Stigma Resistance Text Message Intervention for People Who Use Drugs
Brief Title: Feasibility and Acceptability of a Stigma Text Message Intervention for People Who Use Drugs
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 23-2937; 1F31DA058452 (NIH)
Record Dates: First submitted 2024-02-12; First posted 2024-02-28 (Actual); Results first posted 2024-07-10 (Actual); Last update posted 2024-07-10 (Actual); Status verified 2024-02

CONDITIONS: Stigma, Social; Substance Use
Keywords: people who use drugs; rural health; stigma; behavioral interventions; mobile health; mental health
MeSH Terms: conditions — Social Stigma; Substance-Related Disorders; Psychological Well-Being

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention arm (Experimental): Participants in the intervention arm will receive 56 text messages over 4-weeks.
  Interventions: Behavioral: RESTART

INTERVENTIONS:
Behavioral: RESTART — Project RESTART (Resisting STigma And Revaluating your Thoughts) is a theory-informed, 4-week automated text message intervention to address self-stigma in people who use drugs. The intervention delivers two daily messages to participants for four weeks (56 messages total). Messages address the four components of the personal level of Stigma Resistance Theory: Not believing stigma/catching and challenging stigmatizing thoughts; empowering oneself through learning about substance use and one's own recovery; maintaining one's recovery and proving stigma wrong; and developing a meaningful identity and purpose apart from one's substance use. Content is informed by evidence-based psychotherapeutic approaches (e.g., Acceptance and Commitment Therapy) and health communication theory (e.g., Elaboration Likelihood Model). Messages include psychoeducation about substance use and stigma, coping advice, and suggestions for how to set personal goals, identify values, and build self-esteem.

SUMMARY:
Project RESTART (Resisting STigma And Revaluating your Thoughts) is a theory-informed, 4-week automated text message intervention to address self-stigma in people who use drugs. The intervention delivers two daily messages to participants for four weeks (56 messages total). Messages are designed to address four components of Stigma Resistance Theory: Not believing stigma/catching and challenging stigmatizing thoughts; empowering oneself through learning about substance use and one's own recovery; maintaining one's recovery and proving stigma wrong; and developing a meaningful identity and purpose apart from one's substance use.

This study is a single-group pilot trial to determine whether the intervention is feasible and acceptable to participants. All participants will receive the intervention. The primary outcomes are changes in stigma resistance and self-stigma from baseline to 4-week follow-up using self-report. Implementation and process outcomes will be measured to inform future intervention refinement.

DETAILED DESCRIPTION:
Nearly 850,000 Americans have died from overdose in the past two decades, and mortality reached an all-time high during the COVID-19 pandemic. Substance use disorders (SUD) are more highly stigmatized than other health conditions (e.g., HIV, mental illness). SUD stigma prevents uptake of treatment and harm reduction among people who use drugs (PWUD), contributing to needless morbidity (e.g., infectious disease) and mortality (e.g., overdose), and explains in part why only 6.5% of Americans with SUD received past year treatment. Though key federal agencies have identified stigma as a strategic priority in the epidemic, little is known about how to conceptualize and address SUD stigma compared with other health conditions.

Strategies to address SUD self-stigma, in particular, are severely lacking. Self-stigma manifests in PWUD as internalized stereotypes and fear of experienced stigma, leading to the so-called 'why try' phenomenon in which the stigmatized are disempowered from pursuing life goals. SUD self-stigma is associated with numerous psychosocial outcomes including depression, anxiety, diminished quality of life, maladaptive coping and leads to delays in treatment and harm reduction seeking and retention. To date, SUD interventions have overwhelmingly targeted public stigma such as treatment provider attitudes, while there is a remarkable dearth of evidence-based interventions for addressing self-stigma in PWUD.

Stigma resistance, a coping strategy that promotes resilience through empowerment and positive identity formation, is a promising approach to reducing self-stigma. Stigma resistance is associated with multiple psychosocial outcomes, including reductions in self-stigma and improvements in quality of life, self-efficacy, hope, help-seeking, and recovery. Stigma resistance includes both cognitive and behavioral strategies, such as catching and challenging stigmatizing thoughts, forming positive alternative identities, and empowering oneself through learning about substance use. These strategies align directly with techniques used in the HIV/AIDS and mental illness self-stigma intervention literature. Stigma resistance thus serves as an ideal conceptual framework and menu of strategies for the present study's self-stigma reduction intervention.

Project RESTART (Resisting STigma And Revaluating your Thoughts) is a theory-informed, 4-week automated text message intervention to address self-stigma in people who use drugs. The intervention delivers two daily messages to participants for four weeks (56 messages total). Messages are designed to address four components of Stigma Resistance Theory: Not believing stigma/catching and challenging stigmatizing thoughts; empowering oneself through learning about substance use and one's own recovery; maintaining one's recovery and proving stigma wrong; and developing a meaningful identity and purpose apart from one's substance use.

The specific aim of this study is to evaluate feasibility, acceptability, and preliminary effectiveness of the text message intervention to increase stigma resistance and reduce self-stigma. We will conduct a single-group pilot trial of the intervention among 30 rural Ohio PWUD in active use and collect quantitative and qualitative data at baseline and four-week follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Ages 18 and older at enrollment
* Residing in Scioto County, Ohio at time of enrollment
* Able to speak and read English
* Reliable daily access to smart phone with a data plan capable of sending and receiving text messages during the intervention period (4 weeks)
* Self-reported past 30-day use of illicit opioids (e.g., heroin, fentanyl), prescription opioids not as prescribed (e.g., oxycodone, buprenorphine), methamphetamine, or cocaine
* Willing to provide informed consent

Exclusion Criteria:

* Unable to be consented due to cognitive impairment
* Planning to move out of the study area during the study period
* Unwilling or unable to comply with protocol requirements
* Currently incarcerated in a correctional facility

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2024-02-29 (Actual); Primary Completion 2024-04-14 (Actual); Study Completion 2024-04-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Adams L Sibley, MPH, Principal Investigator — Doctoral Candidate
Locations (1):
- SHRPS Syringe Service Program, Portsmouth, Ohio, United States

IPD SHARING:
Plan to Share IPD: Yes
All of the individual participant data collected during the trial, after deidentification, may be provided to researchers who provide a methodologically sound proposal to achieve the proposal's aims.
Supporting Information: Study Protocol, SAP, ICF, Analytic Code
Time Frame: beginning 9 and continuing for 36 months following publication
Access Criteria: Deidentified individual data that supports the results will be shared beginning 9 to 36 months following publication provided the investigator who proposes to use the data has approval from an Institutional Review Board (IRB), Independent Ethics Committee (IEC), or Research Ethics Board (REB), as applicable, and executes a data use/sharing agreement with UNC. Requests should be submitted via email to the Principal Investigator at asibley@live.unc.edu.

REFERENCES:
- [Derived] Sibley AL, Muessig KE, Noar SM, Gottfredson O'Shea N, Miller WC, Go VF. Promoting substance use stigma resistance through an automated text message intervention (project RESTART): Outcomes of a pilot feasibility trial. J Subst Use Addict Treat. 2025 May;172:209671. doi: 10.1016/j.josat.2025.209671. Epub 2025 Mar 6. PMID 40057241
- [Derived] Sibley AL, Noar SM, Muessig KE, O'Shea NG, Paquette CE, Spears AG, Miller WC, Go VF. An Automated Text Messaging Intervention to Reduce Substance Use Self-Stigma (Project RESTART): Protocol for a Feasibility and Acceptability Pilot Study. JMIR Res Protoc. 2024 Aug 9;13:e59224. doi: 10.2196/59224. PMID 39121478

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Intervention Arm
Started | 30
Completed | 27
Not Completed | 3
Not completed — Lost to Follow-up | 3

BASELINE CHARACTERISTICS:
Arm/Group | Intervention Arm
Number analyzed (Participants) | 30
Age, Continuous [Mean (Standard Deviation); unit: years] | 37.3 (8.7)
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Gender: Men | 13
  Gender: Women | 17
  Gender: Non-binary / third gender | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 30
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2
  White | 27
  More than one race | 1
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 30
Educational Attainment [Count of Participants; unit: Participants]
  Less than high school diploma | 4
  High school diploma or GED | 15
  Some college but no degree | 10
  Associates degree, trade or technical school | 0
  Bachelors degree, other 4 year college degree, or higher | 1
Employment Status [Count of Participants; unit: Participants]
  Working - full-time | 3
  Working - part-time | 3
  Unemployed | 22
  Not in the labor force | 2
Substance Abuse Self-Stigma Scale [Mean (Standard Deviation); unit: units on a scale] — This is a 40-item Likert-type scale that assesses degree to which participants internalize judgment for their substance use and fear experiencing stigma from others. The scale includes four subscales: self-devaluation (8 items), fear of enacted stigma (9 items), stigma avoidance (13 items), and values disengagement (10 items).
  Total scale score ranges from 40-200, where higher scores reflect higher levels of self-stigma. The self-devaluation, fear of enacted stigma, and stigma avoidance subscales are scored normally, while the values disengagement subscale is reverse scored.
  units on a scale | 124.7 (21.2)
Stigma Resistance Scale [Mean (Standard Deviation); unit: units on a scale] — This is a 20-item Likert-type scale that assesses participants' capacity to resist stigma in five domains (self-other differentiation, personal identity, personal cognitions, peer stigma resistance, public stigma resistance).
  All items are scored such that higher scores reflect greater stigma resistance. Total scale score ranges from 20-100.
  units on a scale | 74.7 (12.8)
Adult Dispositional Hope Scale [Mean (Standard Deviation); unit: units on a scale] — This is a 12-item Likert-type scale that assesses participants' hope (i.e., positive attitude toward the future).
  Total scale score ranges from 12-96, where higher scores indicate greater hope.
  units on a scale | 43.8 (10.1)
Rosenberg Self-Esteem Scale [Mean (Standard Deviation); unit: units on a scale] — This is a 10-item Likert-type scale that assesses participants' self-esteem.
  Total scale score range from 10-40, where higher scores indicate greater self-esteem.
  units on a scale | 23.5 (4.5)

OUTCOME MEASURES:

1. Primary Outcome: Change in Stigma Resistance Scale (SRS) Score
Description: This is a 20-item Likert-type scale that assesses participants' capacity to resist stigma in five domains (self-other differentiation, personal identity, personal cognitions, peer stigma resistance, public stigma resistance).
  All items are scored such that higher scores reflect greater stigma resistance. Total scale score ranges from 20-100.
Time Frame: Baseline, 4-week follow-up visit
Population: Includes participants not lost-to-follow-up with complete data.
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Intervention Arm
Number analyzed (Participants) | 25
score on a scale | 6.28 [1.04 to 11.52]

2. Primary Outcome: Change in Substance Abuse Self-Stigma Scale (SASSS) Score
Description: This is a 40-item Likert-type scale that assesses degree to which participants internalize judgment for their substance use and fear experiencing stigma from others. The scale includes four subscales: self-devaluation (8 items), fear of enacted stigma (9 items), stigma avoidance (13 items), and values disengagement (10 items).
  Total scale score ranges from 40-200, where higher scores reflect higher levels of self-stigma. The self-devaluation, fear of enacted stigma, and stigma avoidance subscales are scored normally, while the values disengagement subscale is reverse scored.
Time Frame: Baseline, 4-week follow-up visit
Population: Includes participants not lost-to-follow-up with complete data.
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Intervention Arm
Number analyzed (Participants) | 19
score on a scale | -14.47 [-26.95 to -2.00]

3. Primary Outcome: Percentage of Prospective Participants Eligible for Participation (Feasibility - Recruitment)
Description: Percentage of potential participants screened for study eligibility who are eligible for participation.
Time Frame: From first recruitment visit to last recruitment visit (up to 4 weeks)
Population: Includes all screened prospective participants
Measure: Number; unit: Percentage of participants
Arm/Group | Intervention Arm
Number analyzed (Participants) | 48
Percentage of participants
  Eligible | 93.8
  Ineligible | 6.3

4. Primary Outcome: Percentage of Prospective Participants Recruited Into Study (Feasibility - Enrollment)
Description: Percentage of potential participants screened for study eligibility who enroll in the study.
Time Frame: From first recruitment visit to last enrollment visit (up to 4 weeks)
Population: Includes eligible prospective participants
Measure: Number; unit: Percentage of participants
Arm/Group | Intervention Arm
Number analyzed (Participants) | 45
Percentage of participants
  Enrolled | 66.7
  Not enrolled | 33.3

5. Primary Outcome: Time to Sample Saturation (Feasibility - Recruitment)
Description: Time in days to enroll the full sample size (n=30), starting from the first recruitment visit
Time Frame: From first recruitment visit to last enrollment visit (up to 4 weeks)
Measure: Number; unit: days
Arm/Group | Intervention Arm
Number analyzed (Participants) | 30
days | 14

6. Primary Outcome: Percentage of Participants Retained in Study (Feasibility - Retention)
Description: Percentage of participants enrolled in the study who are retained through study completion (i.e., complete 4-week follow-up survey).
Time Frame: From first enrollment visit to study completion date (up to 8 weeks)
Measure: Number; unit: Percentage of participants
Arm/Group | Intervention Arm
Number analyzed (Participants) | 30
Percentage of participants
  Retained | 90
  Not retained | 10

7. Primary Outcome: Theoretical Framework of Acceptability (TFA) User Questionnaire Score (Acceptability - User)
Description: This is a 16-item Likert-type questionnaire designed to assess acceptability of the intervention from the participants' perspective along the eight dimensions of the Theoretical Framework of Acceptability: affective attitude, burden, ethicality, intervention coherence, opportunity costs, perceived effectiveness, self-efficacy, and general acceptability.
  Total score ranges from 16-64, with higher scores indicating greater acceptability of the intervention.
Time Frame: 4-week follow-up visit
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention Arm
Number analyzed (Participants) | 27
score on a scale | 56.74 (5.49)

8. Primary Outcome: Percentage of Participants With High Text Message Frequency (Feasibility - User)
Description: Percentage of participants who report "every day" to the 5-point Likert-type survey question "Before the start of this program, how often did you send or receive text messages?"
Time Frame: 4-week follow-up visit
Measure: Number; unit: Percentage of participants
Arm/Group | Intervention Arm
Number analyzed (Participants) | 27
Percentage of participants
  Every day | 74.1
  A few times a week | 18.5
  A few times a month | 7.4
  Less than once a month | 0
  Never | 0

9. Primary Outcome: Percentage of Participants With High Text Messaging Comfort (Feasibility - User)
Description: Percentage of participants who report "very comfortable" or "comfortable" to the 5-point Likert-type survey question "Before the start of this program, how comfortable were you with sending or receiving text messages?"
Time Frame: 4-week follow-up visit
Measure: Number; unit: Percentage of participants
Arm/Group | Intervention Arm
Number analyzed (Participants) | 27
Percentage of participants
  Extremely comfortable | 63.0
  Somewhat comfortable | 11.1
  Neither comfortable nor uncomfortable | 11.1
  Somewhat uncomfortable | 11.1
  Extremely uncomfortable | 3.7

10. Primary Outcome: Percentage of Participants With Cell Phone Device Challenges (Feasibility - User)
Description: Percentage of participants who respond "yes" to the binary survey question "Between the start of the program and now, did you experience any challenges or changes with your phone (e.g., lost, broken) that prevented you from receiving or reading text messages?"
Time Frame: 4-week follow-up visit
Measure: Number; unit: Percentage of participants
Arm/Group | Intervention Arm
Number analyzed (Participants) | 27
Percentage of participants
  Yes | 37.0
  No | 59.3
  Unsure | 3.7

11. Primary Outcome: Percentage of Participants With Cell Phone Plan Challenges (Feasibility - User)
Description: Percentage of participants who respond "yes" to the binary survey question "Between the start of the program and now, did you experience any challenges or changes with your phone number or phone plan (e.g., changed number, ran out of minutes) that prevented you from receiving or reading text messages?"
Time Frame: 4-week follow-up visit
Measure: Number; unit: Percentage of participants
Arm/Group | Intervention Arm
Number analyzed (Participants) | 27
Percentage of participants
  Yes | 22.2
  No | 70.4
  Unsure | 7.4

12. Primary Outcome: Percentage of Participants Who Read Messages Daily (Feasibility - User)
Description: Percentage of participants who respond "As soon as I saw them" or "Later that day" to the 5-point Likert-type survey question "On average, when would you read the text message you received?"
Time Frame: 4-week follow-up visit
Measure: Number; unit: Percentage of participants
Arm/Group | Intervention Arm
Number analyzed (Participants) | 27
Percentage of participants
  "As soon as I saw them" or "Later that day" | 100
  "Later that week," "more than one week later," or "Never" | 0

13. Secondary Outcome: Change in Adult Dispositional Hope Scale Score
Description: This is a 12-item Likert-type scale that assesses participants' hope (i.e., positive attitude toward the future).
  Total scale score ranges from 12-96, where higher scores indicate greater hope.
Time Frame: Baseline, 4-week follow-up visit
Population: Includes participants not lost-to-follow-up with complete data.
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Intervention Arm
Number analyzed (Participants) | 24
score on a scale | 1.58 [-2.36 to 5.53]

14. Secondary Outcome: Change in Rosenberg Self-Esteem Scale Score
Description: This is a 10-item Likert-type scale that assesses participants' self-esteem.
  Total scale score range from 10-40, where higher scores indicate greater self-esteem.
Time Frame: Baseline, 4-week follow-up visit
Population: Includes participants not lost-to-follow-up with complete data.
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Intervention Arm
Number analyzed (Participants) | 24
score on a scale | 3.13 [0.41 to 5.84]

ADVERSE EVENTS:
Time Frame: From the time of signing informed consent, through study completion, a total of 1 month.
Arm/Group | Intervention Arm
All-Cause Mortality (participants affected / at risk) | 0/30
Serious Adverse Events (participants affected / at risk) | 0/30
Other Adverse Events (participants affected / at risk) | 0/30

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2024-02-19): https://cdn.clinicaltrials.gov/large-docs/48/NCT06281548/Prot_SAP_001.pdf
  • Informed Consent Form (2024-02-19): https://cdn.clinicaltrials.gov/large-docs/48/NCT06281548/ICF_002.pdf